CLINICAL TRIAL: NCT00280423
Title: A 28 Day, Polysomnographic and Subjective Assessment of GW679769 for the Treatment of Primary Insomnia: A Randomized, Double-blind, Parallel-Group, Placebo-Controlled Trial.
Brief Title: Effects Of GW679769 On Sleep Onset And Maintenance And Next Day Functioning In Subjects With Primary Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAD103894
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Sleep Initiation and Maintenance Disorders; Insomnia
Keywords: Cognition; Polysomnography; Primary Insomnia; Electroencephalography; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — casopitant

INTERVENTIONS:
Drug: GW679769

SUMMARY:
This study is designed to find the optimal (best) doses of GW679769 that could be given daily to promote sleep onset and maintain sleep during the night without significant next-day thinking impairment and drowsiness in subjects with primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Difficulty going to sleep and/or staying asleep for at least the past 3 months.
* Insomnia must result in significant distress or impairment in functioning at home, socially or at work.
* Otherwise good health with no significant or unstable medical disorder including psychiatric, neurological, endocrine, heart, lung or gastrointestinal disorders, drug/alcohol abuse, cognitive impairment, cancer or chronic pain conditions such as arthritis.

Exclusion Criteria:

* History of other sleep disorders such as sleep apnea or restless leg syndrome.
* Regular sleep habits, including bedtime between 9 PM and midnight.
* No nightshift/rotating shift work, frequent napping or planned travel across >2 time zones.
* Use of nicotine, caffeine and alcoholic products.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 342 (Actual)
Dates: Start 2006-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Comparison of GW679769 and placebo on the time needed to fall asleep at bedtime on Nights 1/2, 13/14 and 27/28 of treatment, as assessed by electroencephalography and other physiological changes during sleep. | 28 Days

SECONDARY OUTCOMES:
Comparison of GW679769 and placebo effects on sleep maintenance and duration on Nights 1/2, 13/14 and 27/28 of treatment, as assessed by electroencephalography and subject diaries, and on next-day memory, alertness and physical coordination. | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (60):
- United States (53):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, National City, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Delray Beach, Florida
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Hinesville, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Crestview Hills, Kentucky
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Newton, Massachusetts
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, Hattiesburg, Mississippi
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Clementon, New Jersey
  - GSK Investigational Site, West Seneca, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Beachwood, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Gallipolis, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Gresham, Oregon
  - GSK Investigational Site, Clarks Summit, Pennsylvania
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, Salt Lake City, Utah
- Canada (7):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Niagara Falls, Ontario
  - GSK Investigational Site, Parrry Sound, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec